CLINICAL TRIAL: NCT02317263
Title: A Trial to Investigate the Effectiveness of Testosterone Treatment in Men With Multiple Sclerosis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: NIH did not fund the study so it never started
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01NS089369
Record Dates: First submitted 2014-12-03; First posted 2014-12-15 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-08

CONDITIONS: Multiple Sclerosis
Keywords: MS
MeSH Terms: conditions — Multiple Sclerosis | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testosterone gel (Active Comparator): Apply gel once a day for 96 weeks
  Interventions: Drug: testosterone
- Placebo gel (Placebo Comparator): Apply gel once a day for 96 weeks
  Interventions: Drug: placebo gel

INTERVENTIONS:
Drug: testosterone
  Arms: Testosterone gel
Drug: placebo gel
  Arms: Placebo gel

SUMMARY:
This is a multicenter, prospective, placebo-controlled, double-blind randomized Phase II clinical trial assessing the effect of testosterone treatment vs. placebo treatment for 96 weeks duration on whole brain atrophy in men with MS.

ELIGIBILITY:
Inclusion Criteria: Men, aged 18-60, with a diagnosis of multiple sclerosis by 2010 revised McDonald Criteria

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2099-01 (Estimated); Study Completion 2099-01 (Estimated)

PRIMARY OUTCOMES:
Whole Brain Atrophy | 96 weeks